CLINICAL TRIAL: NCT05124145
Title: Primary Care in AURA for Covid-19: Implementation of a Regional Practice-based Surveillance Network
Brief Title: Primary Care in AURA for COVID-19
Acronym: SOPRAC
Status: Completed | Type: Observational
Sponsor: Research on Healthcare Performance Lab U1290 (Other)
Responsible Party: Sponsor
Other Study IDs: SOPRAC
Record Dates: First submitted 2021-11-16; First posted 2021-11-17 (Actual); Last update posted 2021-11-26 (Actual); Status verified 2021-11

CONDITIONS: Primary Care : Suspected and Confirmed Cases of COVID-19; Primary Health Care; COVID-19 Pandemic
Keywords: COVID-19; Primary care; Clinical epidemiology; Practice assessment
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- surveillance network: The surveillance network is made of 200 health professionals from 85 practices
  Interventions: Other: No intervention (surveillance system)

INTERVENTIONS:
Other: No intervention (surveillance system) — The surveillance network will collect data on all consecutive COVID-19 cases

SUMMARY:
As few data are available on the epidemiology of the COVID-19 in primary care, the project aims to implement a practice-based surveillance network based on multiprofessional health homes in the French region Auvergne-Rhône-Alpes (Aura), able to monitor the evolution of the current epidemic.

ELIGIBILITY:
Inclusion Criteria:

* Suspect or confirmed COVID-19 case consulting in primary care in the Aura region

Exclusion Criteria:

* Patient with a COVID-19 diagnosis excluded after clinical examination or investigation.
* Patient refusing to participate to the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients consulting a health professional in primary care in the AURA region, by physical encounter, visio-consultation or telephone call, during the COVID-19 epidemics period
Sampling Method: Non-Probability Sample
Enrollment: 7000 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2020-11-02 (Actual); Study Completion 2021-11-05 (Actual)

PRIMARY OUTCOMES:
Estimation of the weekly incidence of COVID-19 confirmed cases | 30 days after the COVID-19 suspected
  Confirmed cases will be defined by the positivity of the detection of SARS-CoV-2 in RT-PCR and possibly by serology (for patients in whom a test is performed).
  The incidence rate of confirmed cases will be estimated from the number of new cases confirmed by a positive biological test reported in the patient population of the participating facilities.

CONTACTS AND LOCATIONS:
Overall Officials: Laurent LETRILLART, MD, PhD, Principal Investigator — Research on Healthcare Performance Lab U1290
Locations (1):
- RESHAPE, Lyon, France